CLINICAL TRIAL: NCT06168968
Title: Multidisciplinary Approach to Reduce Cardiovascular Health Disparities in the Baltimore RAcial Minority CommunitiEs (M-BRACE Trial)
Brief Title: Multidisciplinary Approach to Reduce Cardiovascular Health Disparities
Acronym: M-BRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Paul A. Gurbel, Director of Cardiovascular Research, LifeBridge Health
Other Study IDs: 1941089
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome; Multi Vessel Coronary Artery Disease; Ischemic Stroke
MeSH Terms: conditions — Acute Coronary Syndrome; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient: (Secondary Prevention) Includes black (n=150) and white (n=150) patients greater than or equal to 18 years of age hospitalized for acute coronary syndrome (ACS), multi-vessel disease, or ischemic stroke undergoing intervention
  Interventions: Behavioral: Life and Medication Recommendations
- Family Member: (Primary Prevention) Includes black subjects (n=75) who are first or second-degree relatives of patients in Cohort 1 and have no history of prior hospitalization for cardiovascular or cerebrovascular disease
  Interventions: Behavioral: Life and Medication Recommendations

INTERVENTIONS:
Behavioral: Life and Medication Recommendations — Based on obtained subjective and objective data from patient-filled questionnaire and laboratory testing respectively, lifestyle and medication recommendations will be provided for secondary prevention of cardiovascular and cerebrovascular diseases

SUMMARY:
The goal of this observational study is to investigate the potential differences in thrombogenicity between black and white patients admitted with atherothrombotic events including acute coronary syndrome, multi-vessel coronary disease, and ischemic stroke.

Participants will engage in laboratory testing and health outcome assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age admitted with ACS, AIS, or multi-vessel CAD
* Competent mental condition to provide informed consent and able to participate in follow-ups

Exclusion Criteria:

* Pregnant women
* Currently enrolled in an investigational drug or device trial
* Undergoing treatment for neoplastic, autoimmune, or connective tissue disease
* COVID-19 infection within 30 days of enrollment
* Known history of hepatitis or HIV
* Deemed unfit to participate according to the investigator
* Known history of drug abuse
* Known platelet count of <100,000/mm3
* Hematocrit < 25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two Cohorts (Cohort 1 = Secondary Prevention, Cohort 2 = Primary Prevention)
  - See information about specific Cohorts
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences in Platelet Fibrin Clot Formation (MA,mm) | Baseline
  Differences in Platelet Fibrin Clot Formation (MA,mm) Between Black and White Patients
Differences in Speed of Clot Formation (R, min) | Baseline
  Differences in Speed of Clot Formation (R, min) Between Black and White Patients

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events Post Index Hospitalization | 3 and 12 months post index hospitalization
  Major Adverse Cardiovascular Events (death, MI, stroke, unplanned target vessel revascularization, major bleeding) Post Index Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Brager, PhD, Study Chair — LifeBridge Health
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No